CLINICAL TRIAL: NCT05554120
Title: The Next Step in Smoking Prevention: the Reduction of Tobacco Retail Outlets, a Comprehensive Policy Evaluation
Status: Enrolling by invitation | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Investigative Desk (Unknown); SEO Amsterdam Economics (Unknown); IVO Research Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: KWF140282021-2
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-06

CONDITIONS: Smoking, Tobacco; Smoking Behaviors; Smoking Cessation; Smoking Reduction
Keywords: Tobacco; Policy evaluation; Social class; Supermarkets
MeSH Terms: conditions — Tobacco Smoking; Smoking; Smoking Cessation; Smoking Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-smoking adolescents: Non-smoking youth aged 12-17 years old. As the investigators monitor the cohort, it is possible that some of the cohort will become smokers.
  Interventions: Other: Supermarket tobacco sales ban
- Smoking adults from disadvantaged neighbourhoods: Smoking adults aged 18 years and older from disadvantaged neighbourhoods. The investigators distinguish between disadvantaged and non-disadvantaged neighborhoods by using data from CBS Statistics Netherlands (CBS).
  Interventions: Other: Supermarket tobacco sales ban
- Smoking adults from non-disadvantaged neighbourhoods: Smoking adults aged 18 years and older from non-disadvantaged neighbourhoods. The investigators distinguish between disadvantaged and non-disadvantaged neighborhoods by using data from CBS Statistics Netherlands (CBS).
  Interventions: Other: Supermarket tobacco sales ban

INTERVENTIONS:
Other: Supermarket tobacco sales ban — In 2024, a ban on the sales of tobacco for supermarkets is planned by the Dutch government. Supermarkets accounted for approximately 40% of tobacco outlets in the Netherlands in 2021.

SUMMARY:
Few countries have legislation to reduce the number and types of tobacco retail outlets. The Netherlands plans to ban tobacco sales in supermarkets in 2024. The overall aim of this proposed research is to evaluate the implementation of new legislation to reduce the number and types of tobacco outlets in the Netherlands, up until and including the ban on sales of tobacco in supermarkets.

In a comprehensive policy evaluation, the investigators plan to examine (1) the impact of the policy on the number and types of tobacco outlets, (2) the impact on attitudes and behaviors of smoking adults and non-smoking youth, and (3) the influence of the tobacco industry on the policy process and the retail environment. In addition, the investigators plan to focus on differential effects in disadvantaged neighborhoods, where both smoking rates and tobacco outlet density are typically highest.

The investigators bring together a unique combination of economic, psychological, and journalistic research methods. The investigators examine the impact of the new legislation on the amount and type of tobacco outlets and on the number of smokers by using routinely collected monitoring data. The investigators examine the impact of the legislation on smoking susceptibility of non-smoking youth and on impulse tobacco purchases by smoking adults with yearly quantitative surveys (two surveys before the policy implementation and two after) and with qualitative interviews and discussion sessions. The investigators examine whether these impacts differ for disadvantaged versus non-disadvantaged neighborhoods. The investigators examine what strategies the tobacco industry uses to influence the new legislation, policy processes, and the tobacco retail environment by performing a journalistic investigation, using for example documents obtained by Freedom of Information Act requests, (possibly) leaked documents from insider meetings, and interviews with insiders.

Our research will provide a comprehensive evaluation of the effects of the implementation of the proposed legislative measures. Based on our results, the investigators will formulate recommendations for the Dutch Cancer Society, the Dutch government, and for other countries who consider reducing the number of tobacco outlets; highlight potential areas for further development and improvement within the legislative framework and provide recommendations on how to counter the lobby from the tobacco industry.

DETAILED DESCRIPTION:
Problem description: Tobacco use is the primary cause of several cancers; among them lung cancer, which is the leading preventable cause of death in the Netherlands. Yet, tobacco use remains high in the Netherlands, with an adult smoking prevalence of 20%, which is even higher in groups with a lower socioeconomic position. Therefore, reducing the smoking prevalence in all groups in society is one of the three priorities in the Dutch National Prevention Agreement. This Agreement was made with the Dutch government and more than 70 societal organizations, including the Dutch Cancer Society. It consists of a range of voluntary agreements and policy measures to reduce smoking prevalence to 5% or less by 2040. Among these measures is the proposal to reduce the number of outlets that sell tobacco. The government has announced a stepwise approach to ban the sales of tobacco products from various types of outlets. The first step is planned for 2022, with a ban on cigarette dispensing machines. This is followed by a ban on the online sale of tobacco in 2023. In 2024, the largest change is planned with a ban on the sales of tobacco for supermarkets, which currently accounts for approximately 40% of tobacco outlets in the Netherlands. The last step is to phase out the sale of tobacco at petrol stations and convenience stores, so that in the end only specialist tobacco shops can sell tobacco products. The reasoning of the Dutch government for this legislation is to protect young (non-)smokers and adult (former) smokers from exposure to tobacco products and with that from the temptation to smoke and to make impulse purchases, ultimately making it easier to quit smoking and less likely to (re-)initiate smoking. It also adds to the denormalization of smoking as it makes tobacco products disappear from common sight. The proposed measures however lack clear goals, such as a target number of tobacco outlets, nor is there any particular attention given to reducing socioeconomic inequalities in smoking through these measures. Moreover, the tobacco industry is known to try to stop, delay, or weaken legislation before it is implemented, and may try to influence the tobacco retail environment.

Research direction: The investigators will do a comprehensive policy evaluation of the new Dutch legislation on tobacco outlets. The investigators examine:

* The effects of the legislation on the number of tobacco sales outlets.
* The effects of the reduced number of sales outlets (if any) on the number of smokers.
* The effects on smoking susceptibility among non-smoking youth.
* The effects on impulse tobacco purchases of smoking adults.
* How these impacts differ for those living in disadvantaged versus non-disadvantaged neighborhoods.
* The strategies that the tobacco industry uses to influence the national legislation on tobacco outlets.
* And the strategies that the tobacco industry uses to influence the tobacco retail environment in the Netherlands.

Aim: The overall aim of this proposed research is to evaluate the implementation of new legislation to reduce the number and types of tobacco outlets in the Netherlands, up until and including the ban on sales of tobacco in supermarkets.

Primary research questions are:

What is the impact of the new legislation on the number and type of tobacco outlets? What is the impact of the new legislation by supermarkets on the number of smokers? What is the impact of the new legislation on smoking susceptibility of non-smoking youth? What is the impact of the new legislation on impulse tobacco purchases by smoking adults? Does this impact differ for smoking adults living in disadvantaged versus non-disadvantaged neighborhoods? What strategies does the tobacco industry use to influence the new legislation and policy processes? What strategies does the tobacco industry use to influence the tobacco retail environment?

Secondary research questions are:

How do non-smoking youth and smoking adults experience the new legislation? To what extent does the new legislation lead to more illegal (online) sales of tobacco and what is the role of the tobacco industry in this? What is the impact of the new legislation on use and marketing of 'reduced risk' products such as electronic cigarettes and heated tobacco?

Expected outcome: Our research will provide a comprehensive evaluation of the effects of the implementation of the proposed measures on the reduction of tobacco outlets. The four organizations that carry out this research have worked closely together in the past on comparable research projects and will ensure that the three parts of the project will come together to provide a comprehensive picture. Based on our results, the investigators will formulate recommendations for the Dutch Cancer Society, the Dutch government, and for other countries who consider reducing the number of tobacco outlets. The investigators will highlight potential areas for further development and improvement within the legislative framework and provide recommendations on how to counter the lobby from the tobacco industry.

Plan of Investigation:

The proposed research consists of three parts:

1. In the first part, the investigators examine the effects of the legislation on the number of tobacco sales outlets. The investigators also study the effects of the reduced number of sales outlets (if any) on the number of smokers. Both are examined separately for disadvantaged and non-disadvantaged neighborhoods. For this work package the investigators rely on existing data on retail locations and smoking prevalence. The investigators use data from 2018 to 2025 to account for existing trends. This part will be carried out by a research institute that specializes in economic analyses (SEO Amsterdam Economic) sand has done previous analyses with sales outlet and smoking prevalence data.
2. In the second part, the investigators examine the effects of the legislation on smoking susceptibility among nonsmoking youth and on impulse tobacco purchases of smoking adults. The investigators also examine how the effects differ for smoking adults living in disadvantaged versus non-disadvantaged neighborhoods. The investigators will conduct yearly, quantitative survey waves from 2022 to 2025 among a cohort of 250 non-smoking youth, 600 smoking adults from disadvantaged neighborhoods, and 600 smoking adults from non-disadvantaged neighborhoods. The investigators will also carry out in-depth qualitative interviews and discussion sessions with non-smoking youth and smoking adults from these three groups. This part will be carried out by a research institute that specializes in mixed-methods addiction research (IVO research Institute) and focuses on vulnerable groups in society, together with a university department of Health Promotion (Maastricht University) that has ample experience with tobacco control policy evaluations.
3. In the third part, the investigators examine the strategies of the tobacco industry to influence both the national legislation on tobacco outlets, and to influence the tobacco retail environment. The investigators use investigative journalism techniques to uncover lobbying strategies and tactics of the tobacco industry and their allies. The investigators use a wide range of sources: documents obtained by FOIA-requests, (possibly) leaked documents from insider meetings, (background) interviews with insiders of the tobacco industry, the government, and the retail sector, the analysis of social media campaigns, financial and marketing data, and observations of tobacco outlets (online and offline). This part will be carried out by an organization of investigative journalists that specializes in the strategies and tactics of the tobacco industry (The Investigative Desk).

ELIGIBILITY:
Group non-smoking adolescents

Inclusion Criteria:

* Dutch-speaking
* aged 12 to 17 years old at enrollment

Exclusion Criteria:

* they have smoked (part of) a cigarette at least once a month during the last six months
* not providing informed consent to participate

Smoking adults

Inclusion Criteria:

* Dutch-speaking
* smoking at least monthly at enrollment
* having smoked at least 100 cigarettes in their lifetime

Exclusion Criteria:

* not providing informed consent to participate

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Respondents are recruited from NIPObase, a large probability-based access database that mirrors the Dutch population. NIPObase includes over 103,000 respondents in the general population who regularly participate in surveys from Kantar. With NIPObase the investigators are able to draw samples that are representative of the Dutch population according to known characteristics such as gender, age, geographic region, and household size.
Sampling Method: Non-Probability Sample
Enrollment: 1450 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Impulse purchases of tobacco | October 2022; October-November 2023, 2024, 2025
  This is measured amongst smoking adults with the question "When you are shopping in a store in your neighborhood for something other than cigarettes, how often do you decide to buy cigarettes?" (1=Often, 2=Rarely, 3=Sometimes, 4=Often, 5=Always) (Siahpush et al., 2016).
Smoking susceptibility | October 2022; October-November 2023, 2024, 2025
  This is measured amongst non-smoking adolescents with a three-item index, averaging responses to "Would you try smoking a cigarette if one of your best friends offered it to you?", "Do you think you would smoke in the next 6 months?", and "Are you curious about smoking?" (1=Definitely Not, 2=Probably Not, 3=Probably Yes, 4=Definitely Yes) (Strong et al., 2015).
Number of smokers | 2018-2025
  The investigators use data at the individual level. The investigators propose to use existing data from the lifestyle monitor of CBS (15,000 observations annually) and the polling station survey among students (8,000 observations every four years). For each individual the investigators link the area where they live.

SECONDARY OUTCOMES:
Illegal (online) sales of tobacco | October 2022; October-November 2023, 2024, 2025
  The investigators will ask our adult cohort if they have "bought cigarettes or tobacco during the past 6 months from people who sell cigarettes or tobacco independently, for example at the door or on the street" and the frequency of which they do so.
  The investigators will also do observations on the Internet, for mapping the developments in (online) sales, possibly also via 'scraping'. This technique involves systematically gathering and arranging data from a large number of websites and provides insight into the development of the number of (online) sales sites, of product pricing, of changes in product availability and of the overall 'traffic' (visitor amount) of these websites, indicating (legal or illegal) shopping activities.
Use and marketing of 'reduced risk' products | October 2022; October-November 2023, 2024, 2025
  The investigators adopt a wide definition of 'reduced risk' products. The use of the products will be measured in our cohort and with investigative journalism methods. Marketing of the products will also be explored with investigative journalism methods.
Number and type of tobacco outlets | 2018-2025
  For the number and type of tobacco outlets the investigators rely on existing data from Locatus. Locatus is a company which collects information about retail locations on a daily basis by professional field service.
  They can distinguish the following types of outlets:
  * Supermarkets
  * Mini supermarkets
  * Petrol stations (staffed)
  * Convenience stores: they sell tobacco and convenience articles like journals, lottery tickets, office supplies, greeting cards, telephone accessories and candies
  * Specialist tobacco shops (with more than 70% of turnover from tobacco sales)
  * Night shops.

CONTACTS AND LOCATIONS:
Overall Officials: Gera E Nagelhout, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siahpush M, Shaikh RA, Hyland A, Smith D, Sikora Kessler A, Meza J, Wan N, Wakefield M. Point-of-Sale Cigarette Marketing, Urge to Buy Cigarettes, and Impulse Purchases of Cigarettes: Results From a Population-Based Survey. Nicotine Tob Res. 2016 May;18(5):1357-62. doi: 10.1093/ntr/ntv181. Epub 2015 Sep 16. PMID 26377520
- [Background] Strong DR, Hartman SJ, Nodora J, Messer K, James L, White M, Portnoy DB, Choiniere CJ, Vullo GC, Pierce J. Predictive Validity of the Expanded Susceptibility to Smoke Index. Nicotine Tob Res. 2015 Jul;17(7):862-9. doi: 10.1093/ntr/ntu254. Epub 2014 Dec 6. PMID 25481915
- [Derived] Nagelhout GE, Poole NL, Metze M, Willemsen MC, Vermeulen W, van den Brand FA. Reducing the number and types of tobacco retail outlets in the Netherlands: Study protocol for a comprehensive mixedmethods policy evaluation. Tob Prev Cessat. 2023 Mar 29;9:08. doi: 10.18332/tpc/161825. eCollection 2023. PMID 37009236